CLINICAL TRIAL: NCT04712526
Title: Safety and Efficacy of the AEON™ Endostapler in Laparoscopic Roux-en-Y Gastric Bypass Surgery
Brief Title: Endostapler Gastric Bypass Study
Status: Withdrawn | Type: Observational
Why Stopped: voluntarily withdrawn
Sponsor: Lexington Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Endostapler03
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- AEON Endostapler: Stapling performed with AEON Endostapler
  Interventions: Device: AEON Endostapler

INTERVENTIONS:
Device: AEON Endostapler — Surgery with AEON Endostapler

SUMMARY:
The goal of this prospective, post-market study is to evaluate safety and efficacy of the AEON™ Endostapler when used in laparoscopic Roux-en-Y gastric bypass surgery.

DETAILED DESCRIPTION:
Stapler performance will be evaluated by incidence and degree of staple line bleeding from endoscopic and laparoscopic images, evaluated by a third-party. The study will include 25 total consecutive cases of individuals undergoing a planned laparoscopic Roux-en-Y gastric bypass (GB). The GB procedure will be performed according to institutional standard-of-care and all subjects will undergo standard preoperative evaluation as well as post-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned laparoscopic Roux-en-Y gastric bypass
* Informed consent for study obtained and signed from each subject

Exclusion Criteria:

* Planned open surgical approach
* Use of staple line reinforcement material (buttress)
* Revision or other bariatric procedure
* Patients with a bleeding disorder: known coagulopathy, or Platelets <100,000, or PTT > 45sec, or PT> 15sec, or INR>1.5
* Patients with active HIV or Hepatitis B
* Patients under the age of 18 on the date of the surgery
* Patients who are pregnant
* Patients using tobacco products within the last 2 weeks prior to surgery date
* Patients using cortisone or related products within the last 2 weeks prior to surgery date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of reported device-related adverse events | Within 30-day post-operative period

SECONDARY OUTCOMES:
Endoscopic staple line bleeding | Within surgery
  Incidence of intraoperative staple line bleeding from endoscopic images as measured by the provided bleeding severity scale - Bleeding Severity Scale for Endoscope Images (1: No bleeding, 5: Profuse Bleeding)
Laparoscopic staple line bleeding | Within surgery
  Incidence of intraoperative staple line bleeding from laparoscopic images as measured by the provided bleeding severity scale - Bleeding Severity Scale for Laparoscope Images (1: No bleeding, 5: Profuse Bleeding)
Incidence of intraoperative or postoperative blood transfusion | Within 72 hours of surgery start time
Incidence of product malfunction | Within surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Holyoke Medical Center, Holyoke, Massachusetts, United States